CLINICAL TRIAL: NCT05500079
Title: Efficacy of Transctunaous Pulsed Radiofrequency Therapy in Carpal Tunnel Syndrome
Brief Title: Transctunaous Pulsed Radiofrequency Therapy in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Director, medical doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Carpal Tunnel Syndrome
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Neuropathy; Chronic Pain
Keywords: carpal tunnel syndrome; pulsed radiofrequency treatment; transcutaneous pulsed radiofrequency
MeSH Terms: conditions — Peripheral Nervous System Diseases; Chronic Pain; Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wrist splint group (Active Comparator): The group to be treated with a wrist splint
  Interventions: Device: Wrist splint
- Transcutaneous pulsed RF group (Active Comparator): The group to be treated with transcutaneous pulsed RF
  Interventions: Other: Pulsed radiofrequency current

INTERVENTIONS:
Device: Wrist splint — A wrist splint is a It stabilizes your wrist. Wearing a wrist splint minimizes pressure on the median nerve.
  Arms: Wrist splint group
Other: Pulsed radiofrequency current — Pulsed rf current is delivered to the median nerve trace via transcutaneous pads. Pain expression is suppressed in the dorsal horn of the spinal cord.
  Arms: Transcutaneous pulsed RF group

SUMMARY:
The aim of this study is to examine the effect of transcutaneous pulsed radiofrequency current in the treatment of carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common peripheral neuropathy. Wrist splint is the first-line treatment option for CTS. Pulsed radiofrequency therapy is used in the treatment of chronic pain.

60 carpal tunnel syndrome patients diagnosed with electroneuromyelography will be included in the study. 30 patients will wear wrist splints for 1 month. In the other 30 patients, pulsed radiofrequency current will be given through the wrist median nerve trace. RF current will be applied through transcutaneous pads. It will be applied once a week for a total of 2 sessions, 8 minutes each. Boston carpal tunnel syndrome questionnaire with visual analog scale (VAS) will be applied to all patients before and after the treatment at 1 week and 1 month.

Our aim is to compare the effectiveness of wrist splint and pulsed rf therapy.

ELIGIBILITY:
Inclusion Criteria:

* Carpal tunnel syndrome detected by electroneuromyography
* Positive Tinel sign

Exclusion Criteria:

* Thenar muscle atrophy
* Weakness in the abductor pollicis brevis muscle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain on the Visual Analog Scale (VAS) at Week 2 and 4 | Baseline, Week 2 and 4
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "0=no pain" and "10=worst pain.
Boston Carpal Tunnel Syndrome Questionnaire before treatment | Before treatment
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a disease-specific measure of self-reported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome.
  ıncluding Symptom Severity Scale is 11: no symptoms, 55: worst symptoms and Functional Disability Scale (FDS) no difficulties:8, worst difficulties: 40

CONTACTS AND LOCATIONS:
Overall Officials: mehlika panpallı ateş, Study Chair — Diskapi TRH; ömer taylan akkaya, Study Director — Diskapi TRH; Hüseyin Alp Alptekin, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Yildirim Beyazıt Teaching and Research Hospital, Ankara, Dişkapi, Turkey (Türkiye)